CLINICAL TRIAL: NCT07063576
Title: Effect of Baclofen as an Add on Therapy in Management of Patients With Gastroesophageal Reflux Disease Symptoms
Brief Title: Effect of Baclofen in Management of Patients With Gastroesophageal Reflux Disease Symptoms
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Adnan Imtiaj Rahul (Other)
Responsible Party: Sponsor-Investigator, Adnan Imtiaj Rahul, Principal investigator, Dhaka Medical College
Organization: Dhaka Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-DMC/2025/70
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: GERD - PPI Non-responders
Keywords: baclofen; GERD symptoms
MeSH Terms: interventions — Baclofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baclofen (Active Comparator): Tablet baclofen 10mg three times will be given along with conventional treatment
  Interventions: Drug: Baclofen 10mg
- Placebo (Placebo Comparator): Tablet placebo three times daily along with conventional treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baclofen 10mg — Tablet baclofen 10mg three times daily along with conventional treatment
  Arms: Baclofen
Drug: Placebo — Tablet placebo three times daily along with conventional treatment
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the effect of using baclofen along with conventional treatment in improving GERD symptoms. It will also assess the safety of drug baclofen by recording the patient reported adverse events. The main questions it aims to answer are :

Does drug baclofen along with conventional treatment has any effect on patients with GERD symptoms? What medical problems do participants have when taking drug baclofen? Researcher will compare drug baclofen along with conventional treatment to a control group taking placebo along with conventional treatment.

Participants will:

Take drug baclofen 10 milligrams or placebo three times daily along with conventional treatment for 4 weeks. They will visit the hospital after 4 weeks. Their symptoms will be assessed via validated GERD Q questionnaire at baseline and after 4 weeks. Additionally, patient reported adverse events will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* Patients with persistent GERD symptoms (Heart burn and/or regurgitation) despite taking conventional treatment including PPI for 8 weeks

Exclusion Criteria:

* GERD symptoms with any alarming features (dysphagia, weight loss, bleeding, vomiting, and/or anemia)
* Baseline GERD Q score less than 8
* Peptic gastric or duodenal ulcer on endoscopy
* Other esophageal disease like achalasia, carcinoma, corrosive stricture
* Gastrointestinal malignancy
* History of major gastrointestinal surgery
* Medical disease that affects the esophageal or gastric motility, such as uncontrolled diabetes, hyperthyroidism, hypothyroidism
* Patient with renal impairment
* Pregnant and lactating women
* Use of drugs affecting on LES
* Regular use of drug that may interact with Baclofen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of GERD symptoms | At baseline before randomization and at week 4
  The improvement of GERD symptoms will be assessed by GERD Q questionnaire.

SECONDARY OUTCOMES:
Effect of baclofen along with conventional treatment | At week 4
  Effect of baclofen along with conventional treatment including PPI on GERD symptoms will be assessed by GERD Q questionnaire
Effect of placebo along with conventional treatment | At 4 week
  Effect of placebo along with conventional treatment including PPI on GERD symptoms will be assessed by GERD Q questionnaire
Comparison of effects of baclofen and placebo along with conventional treatment | At week 4
  Comparison of effects of baclofen and placebo along with conventional treatment including PPI on GERD symptoms will be assessed by GERD Q questionnaire
Adverse events | Through the completion of study approximately one year
  Patients reported adverse events will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh